CLINICAL TRIAL: NCT00983983
Title: Phase II Safety and Tolerability Study of High Fat/High Calorie Versus High Calorie Versus Optimal Nutrition in Subjects With Amyotrophic Lateral Sclerosis
Brief Title: High Fat/High Calorie Trial in Amyotrophic Lateral Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Muscular Dystrophy Association (Other)
Responsible Party: Principal Investigator, Anne-Marie Alexandra Wills, MD, Assistant Professor of Neurology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MDA136152; 2009-P-001132
Record Dates: First submitted 2009-09-23; First posted 2009-09-24 (Estimated); Results first posted 2015-02-27 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2015-02

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; ALS; Motor Neuron Disease; MND; Fat; Lipid; Cholesterol; Omega-3 fatty acid; Diet; Tube feed; Gastrostomy; PEG; Adults with Amyotrophic Lateral Sclerosis (ALS)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease; Platelet Glycoprotein IV Deficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High fat/high calorie (Experimental): High fat/high calorie diet: Oxepa
  Interventions: Dietary Supplement: Oxepa
- High calorie (Active Comparator): High calorie diet: Jevity 1.5
  Interventions: Dietary Supplement: Jevity 1.5
- Control (Placebo Comparator): Control diet: Jevity 1.0
  Interventions: Dietary Supplement: Jevity 1.0

INTERVENTIONS:
Dietary Supplement: Oxepa — Oxepa: Tube feed containing 1.5 calories/ml of which 55% calories are from fat, including eicosapentaenoic acid and gamma-linolenic acid. Subjects will receive 1.25 times their daily caloric requirements based on their measured resting energy expenditure. Subjects will receive 4 months of tube feeds and be followed for an additional 1 month to measure adverse events and tolerability.
  Arms: High fat/high calorie
Dietary Supplement: Jevity 1.5 — Jevity 1.5: Tube feed containing 1.5 calories/ml of which 29.4% are from fat. Subjects will receive 1.25 times their daily caloric requirements based on their measured resting energy expenditure. Subjects will receive 4 months of tube feeds and be followed for an additional 1 month to measure adverse events and tolerability.
  Arms: High calorie
Dietary Supplement: Jevity 1.0 — Jevity 1.0: Control tube feed. Subjects will receive 1.0 times their daily caloric requirements based on their measured resting energy expenditure. Subjects will receive 4 months of tube feeds and be followed for an additional 1 month to measure adverse events and tolerability.
  Arms: Control

SUMMARY:
The purpose of this study is to determine the safety, tolerability, and preliminary efficacy of long-term use of high fat/high calorie and high calorie diets in people with amyotrophic lateral sclerosis (ALS) (Lou Gehrig's disease).

DETAILED DESCRIPTION:
Weight loss is a common and severe symptom of amyotrophic lateral sclerosis (ALS), caused both from inadequate calorie intake and an increased metabolic rate. People with ALS are generally instructed to increase their calorie intake; however, the ideal amount and type of calories has not been studied. Several studies in an animal model of motor neuron disease have shown that a high fat/high calorie diet can increase survival by as much as 38%. Mice on a high fat diet also live longer than mice fed diets consisting of high protein or high sugar. We are therefore conducting a phase II safety, tolerability, and preliminary efficacy trial in ALS of high fat versus high calorie versus normal diet. The normal diet will be calculated based on the number of calories needed to replace each participant's measured daily calorie requirement.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of ALS
2. Male or female subjects aged 18 years or older
3. Must already be tolerating tube feedings through either a gastrostomy tube (G-tube or PEG) or jejunostomy tube (J-tube)
4. Must require non-invasive ventilation (BIPAP) for less than 10 hours/day
5. Women of childbearing potential must have a negative pregnancy test at screening and be non-lactating.

Exclusion Criteria:

1. History of hepatitis including non-alcoholic steatohepatitis (NASH), cholecystectomy, prior biliary disease such as gallstones
2. History of diabetes
3. History of prior myocardial infarction or stroke
4. Laboratory values: Screening alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than 2.0 times the upper limit of normal or total bilirubin greater than 1.5 times the upper limit of normal
5. Allergy to soy, fish, or milk products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-10; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Marie A Wills, M.D., Principal Investigator — Massachusetts General Hospital
Locations (13):
- United States (13):
  - Barrow Neurological Institute/St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - University of California at Irvine, Irvine, California
  - California Pacific Medical Center, University of California at San Francisco, San Francisco, California
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Neurology Clinical Trials Unit, Massachusetts General Hospital, Boston, Massachusetts
  - Saint Mary's Health Care, Grand Rapids, Michigan
  - Columbia Presbyterian Medical Center, New York, New York
  - Carolinas Medical Center Neuromuscular/ALS-MDA Center, Charlotte, North Carolina
  - Oregan Health and Science University, Portland, Oregon
  - Drexel University, Philadelphia, Pennsylvania
  - Methodist Neurological Institute, Houston, Texas
  - University of Vermont, Burlington, Vermont

REFERENCES:
- [Background] Kasarskis EJ, Berryman S, Vanderleest JG, Schneider AR, McClain CJ. Nutritional status of patients with amyotrophic lateral sclerosis: relation to the proximity of death. Am J Clin Nutr. 1996 Jan;63(1):130-7. doi: 10.1093/ajcn/63.1.130. PMID 8604660
- [Background] Desport JC, Torny F, Lacoste M, Preux PM, Couratier P. Hypermetabolism in ALS: correlations with clinical and paraclinical parameters. Neurodegener Dis. 2005;2(3-4):202-7. doi: 10.1159/000089626. PMID 16909026
- [Background] Desport JC, Preux PM, Magy L, Boirie Y, Vallat JM, Beaufrere B, Couratier P. Factors correlated with hypermetabolism in patients with amyotrophic lateral sclerosis. Am J Clin Nutr. 2001 Sep;74(3):328-34. doi: 10.1093/ajcn/74.3.328. PMID 11522556
- [Background] Morozova N, Weisskopf MG, McCullough ML, Munger KL, Calle EE, Thun MJ, Ascherio A. Diet and amyotrophic lateral sclerosis. Epidemiology. 2008 Mar;19(2):324-37. doi: 10.1097/EDE.0b013e3181632c5d. PMID 18300717
- [Background] Veldink JH, Kalmijn S, Groeneveld GJ, Wunderink W, Koster A, de Vries JH, van der Luyt J, Wokke JH, Van den Berg LH. Intake of polyunsaturated fatty acids and vitamin E reduces the risk of developing amyotrophic lateral sclerosis. J Neurol Neurosurg Psychiatry. 2007 Apr;78(4):367-71. doi: 10.1136/jnnp.2005.083378. Epub 2006 Apr 28. PMID 16648143
- [Background] Mattson MP, Cutler RG, Camandola S. Energy intake and amyotrophic lateral sclerosis. Neuromolecular Med. 2007;9(1):17-20. doi: 10.1385/nmm:9:1:17. PMID 17114821
- [Background] Dupuis L, Oudart H, Rene F, Gonzalez de Aguilar JL, Loeffler JP. Evidence for defective energy homeostasis in amyotrophic lateral sclerosis: benefit of a high-energy diet in a transgenic mouse model. Proc Natl Acad Sci U S A. 2004 Jul 27;101(30):11159-64. doi: 10.1073/pnas.0402026101. Epub 2004 Jul 19. PMID 15263088
- [Result] Wills AM, Hubbard J, Macklin EA, Glass J, Tandan R, Simpson EP, Brooks B, Gelinas D, Mitsumoto H, Mozaffar T, Hanes GP, Ladha SS, Heiman-Patterson T, Katz J, Lou JS, Mahoney K, Grasso D, Lawson R, Yu H, Cudkowicz M; MDA Clinical Research Network. Hypercaloric enteral nutrition in patients with amyotrophic lateral sclerosis: a randomised, double-blind, placebo-controlled phase 2 trial. Lancet. 2014 Jun 14;383(9934):2065-2072. doi: 10.1016/S0140-6736(14)60222-1. Epub 2014 Feb 28. PMID 24582471
- [Derived] Paganoni S, Deng J, Jaffa M, Cudkowicz ME, Wills AM. Body mass index, not dyslipidemia, is an independent predictor of survival in amyotrophic lateral sclerosis. Muscle Nerve. 2011 Jul;44(1):20-4. doi: 10.1002/mus.22114. Epub 2011 May 23. PMID 21607987

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 4 participants were screened but excluded due to not meeting inclusion criteria (1 due to history of Myocardial Infarction, 1 due to Diabetes, 1 due to low forced vital capacity, and 1 due to the investigator's judgment).
Period: Overall Study
Arm/Group | High Fat/High Calorie | High Calorie | Control
Started | 8 | 9 | 7
Completed | 6 | 8 | 6
Not Completed | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- High Calorie/High Carbohydrate: High calorie diet: Jevity 1.5
  Jevity 1.5: Jevity 1.5: Tube feed containing 1.5 calories/ml of which 29.4% are from fat. Subjects will receive 1.25 times their daily caloric requirements based on their measured resting energy expenditure. Subjects will receive 4 months of tube feeds and be followed for an additional 1 month to measure adverse events and tolerability.
- Total: Total of all reporting groups
Arm/Group | High Fat/High Calorie | High Calorie/High Carbohydrate | Control | Total
Number analyzed (Participants) | 8 | 9 | 7 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (6.9) | 57.5 (15.4) | 63.2 (9.4) | 61.3 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 1 | 11
  Male | 3 | 4 | 6 | 13
Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) [Mean (Standard Deviation); unit: units on a scale] — Total Score ranging from 0 (worst) to 48 (best)
  units on a scale | 30.7 (7.0) | 25.5 (9.4) | 23.0 (3.5) | 26.3 (7.6)

OUTCOME MEASURES:

1. Secondary Outcome: Rate of Change in ALSFRS-R in Units/Month
Description: Rate of change in the ALS Functional Rating Scale-Revised, calculated in units/month. Negative numbers refer to worsening over time.
Time Frame: Over 5 months
Measure: Mean (95% Confidence Interval); unit: units on a scale/month
Arm/Group | High Fat/High Calorie | High Calorie/High Carbohydrate | Control
Number analyzed (Participants) | 6 | 8 | 6
units on a scale/month | -1.54 [-2.36 to -0.73] | -1.07 [-1.71 to -0.42] | -2.17 [-3.24 to -1.10]
Statistical Analysis 1: Comparison: High Calorie/High Carbohydrate vs Control; Change over time in the ALSFRS-R was analyzed using random-slopes models; Test type: Superiority or Other; p = 0.07, Mixed Models Analysis

2. Secondary Outcome: Biomarkers of Body Composition and Lipid Metabolism
Time Frame: 5 months follow-up
Reporting Status: Not Posted

3. Primary Outcome: Safety Outcomes: Frequency of Adverse Events
Time Frame: 5 months
Measure: Number; unit: Total Number of Adverse Events
Arm/Group | High Fat/High Calorie | High Calorie | Control
Number analyzed (Participants) | 8 | 9 | 7
Total Number of Adverse Events | 49 | 24 | 42
Statistical Analysis 1: Comparison: High Calorie vs Control; Test type: Superiority or Other; p = 0.06, Fisher Exact

4. Primary Outcome: Serious Adverse Events
Description: SAE were defined using the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0.
Time Frame: 5 months
Measure: Number; unit: Number of Serious Adverse Events
Arm/Group | High Fat/High Calorie | High Calorie | Control
Number analyzed (Participants) | 8 | 9 | 7
Number of Serious Adverse Events | 3 | 0 | 9
Statistical Analysis 1: Comparison: High Calorie vs Control; Test type: Superiority or Other; p = 0.0005, Fisher Exact

5. Primary Outcome: Tolerability
Description: Number of participants who completed the study on their assigned study intervention.
Time Frame: 5 months
Population: The number of participants who received the study diet (4 participants withdrew consent prior to receiving study intervention).
Measure: Number; unit: participants
Arm/Group | High Fat/High Calorie | High Calorie | Control
Number analyzed (Participants) | 6 | 8 | 6
participants | 5 | 7 | 1
Statistical Analysis 1: Comparison: High Calorie vs Control; Test type: Superiority or Other; p = 0.03, Fisher Exact

ADVERSE EVENTS:
Time Frame: Participants were followed for adverse events for 30 days after stopping study diet.
Description: Safety analyses were performed on all participants who initiated study diets.
Arm/Group | High Fat/High Calorie | High Calorie/High Carbohydrate | Control
Serious Adverse Events (participants affected / at risk) | 3/6 | 0/8 | 4/6
Other Adverse Events (participants affected / at risk) | 6/6 | 8/8 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Fat/High Calorie (N=6) | High Calorie/High Carbohydrate (N=8) | Control (N=6)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Stomach Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Infection-Lung (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Fat/High Calorie (N=6) | High Calorie/High Carbohydrate (N=8) | Control (N=6)
Allergic Rhinitis (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Elevated Troponin (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1) | 2 (4)
Insomnia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Weight Loss (General disorders) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (4) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 4 (5) | 1 (1) | 3 (3)
Bloating/Flatulence (Gastrointestinal disorders) | 1 (2) | 1 (1) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Detached feeding tube/Replacement of feeding tube (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Heartburn (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Infection-Urinary Tract (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Infection-Bronchus (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (3) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Pain-Abdomen (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Dyspnea-Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 1 (1) | 1 (1)
Cough/Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Pleural Effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Head Cold/Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Sore Throat (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Blocked Foley Catheter (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
"Right arm and leg puffiness" (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Weight Gain (General disorders) | 0 (0) | 1 (1) | 1 (1) — While this was the pre-specified purpose of the study, some sites included this as an AE.
Abrasion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Drooling (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dry Mouth (General disorders) | 1 (1) | 0 (0) | 0 (0)
Esophagitis/Esophageal Spasm (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Burping (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Borborygmi (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Increased Bowel Movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal Fullness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Upset Stomach (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Protein-Calorie Malnutrition (General disorders) | 0 (0) | 0 (0) | 1 (1) — Diagnosed based upon albumin levels during a hospital admission
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Infection-Lung (Pneumonia) (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Oral/Perioral Infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
C. difficile Infection (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Extremity Weakness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Weakness-Trunk (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neck Muscle Soreness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Pain-Abdomen/Stomach (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Pain at PEG site (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No